CLINICAL TRIAL: NCT03290092
Title: A Multi-Centre, Open Label, Single Arm, Phase IB/IIA, Trial of Taselisib (GDC0032) in PIK3CA-Related Overgrowth
Brief Title: Trial of Taselisib in Overgrowth
Acronym: TOTEM
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: In accordance with the protocol, following the occurrence of two SUSARs, the TOTEM trial was stopped early for safety reasons.
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OLIVIER-FAIVRE ROCHE 2016
Record Dates: First submitted 2017-09-19; First posted 2017-09-21 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: PIK3CA-Related Overgrowth
MeSH Terms: interventions — 2-(3-(2-(1-isopropyl-3-methyl-1H-1,2-4-triazol-5-yl)-5,6-dihydrobenzo(f)imidazo(1,2-d)(1,4)oxazepin-9-yl)-1H-pyrazol-1-yl)-2-methylpropanamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Taselisib (GDC0032)

INTERVENTIONS:
Drug: Taselisib (GDC0032) — The first six participants cohort receive a starting dose of 1mg once daily of taselisib during four weeks.
Drug: Taselisib (GDC0032) — The starting dose of the second cohort of 24 patients is 2 mg once daily. This dose may be adjusted down according to the pharmacokinetic data or tolerability data derived from the first cohort.

SUMMARY:
Segmental overgrowth disorders are rare conditions characterised by abnormal growth which is usually asymmetric and confined to discrete parts of the body. We and others have identified mosaic activating mutations in the p110α catalytic subunit of phosphatidylinositol-3-kinase (PI3K; encoded by the PIK3CA gene) in a subset of overgrowth disorders. The PI3K-AKT-mTOR is a critical signalling pathway, which regulates cellular growth, proliferation and survival. Activating mutations in PIK3CA lead to increased activation of the PI3K-AKT-mTORC1 axis, which in turn promotes excessive growth in affected tissue.

The PIK3CA-related overgrowth spectrum is wide, and depends upon the timing of the founder mutation in embryogenesis, and potentially upon the exact mutation. Clinical presentation ranges from isolated enlargement of a digit, to extensive overgrowth of limbs, abdomen and in some cases the brain, and may be accompanied by vascular or lymphatic malformations. Associated morbidity can be profound, with functional impairment, debilitating haemorrhages and thromboses, coupled with neurological sequelae and, in some cases, death. At present, serial debulking surgery is the only available therapeutic option.

The identification of gain-of-function mutations in PI3K has raised the possibility of treatment with drugs that inhibit PIK3CA (the p110 alpha catalytic subunit of PI3K). Taselisib is a selective inhibitor of class I PI3Ks and has direct inhibitory activity of the p110α isoform with a Kiapp value of 0.29 nmol/l.

ELIGIBILITY:
Inclusion Criteria:

* Have given, or their legal representative has given, written informed consent to participate
* Aged 16 years to 65 years inclusive
* Male or female
* Post-zygotic PIK3CA mutation
* Clinically stable in the opinion of the investigator
* Participant Pregnancy and contraception:

  o Female participants of child bearing potential must use an effective method of contraception during treatment and for at least 3 months after the final dose of taselisib. Acceptable methods are:
* True abstinence (this must be the participant's usual and preferred lifestyle, not just for the duration of the trial)
* Oral contraceptive (either combined or progestogen alone)
* Contraceptive implant, injections or patches
* Vaginal ring
* Intrauterine device (IUD, coil or intrauterine system)
* Condom and cap
* Diaphragm plus spermicide

  * A female participant of child bearing potential is defined as a sexually mature woman not surgically sterilized or not post-menopausal for at least 12 consecutive months if aged 55 years or older.
  * Men must use one of the following, reliable forms to contraception for the entire duration of treatment and for 3 months after the final dose of taselisib:
* Condom plus spermicide even if female partner is using another method of contraception (Men should also use a condom to protect male partners, or female partners who are pregnant or breast feeding, from exposure to the Trial medicine in semen).
* True abstinence (this must be the participant's usual and preferred lifestyle, not just for the duration of the Trial)

Exclusion Criteria:

* Pregnant or breastfeeding
* HIV infection
* Hypersensitivity to taselisib or any of its excipients
* Any current medical disorder or medication likely to impair ability to follow the trial protocol safely and effectively
* Are concurrently taking an mTOR inhibitor or any other small molecule inhibitor of the PI3K-AKT signalling pathway
* Unable or unwilling to give informed consent
* Sirolimus or taselisib treatment in 12 weeks prior to screening
* Treatment with a strong inducer or inhibitor of CYP3A4 without the possibility to stop this medication within the week prior to the screening. This includes:
* Macrolide Antibiotics: clarithromycin, telithromycin, erythromycin, troleandomycin
* Gastrointestinal prokinetic agents: metoclopramide.
* Antifungals: itraconazole, ketoconazole, fluconazole, voriconazole, clotrimazole
* Calcium channel blockers: verapamil, diltiazem, nicardipine
* Grapefruit containing foods/drinks
* Anticonvulsants: carbamazepine, phenobarbital, phenytoin
* Antibiotics: rifampicin, rifabutin, rifapentine
* Herbal preparations: St. John's wort (Hypericum perforatum). Other drugs: bromocriptine, cimetidine, danazol, cyclosporine, lansoprazole, calcium containing antacids.
* Inability to attend trial visits
* If less than 3 months post- major surgery at screening
* Any past medical history of inflammatory bowel disease or chronic diarrhoea of unknown aetiology
* History of type 1 or type 2 diabetes mellitus requiring insulin, GLP-1 analogues or oral hypoglycaemic agents.
* History of inflammatory bowel disease, ischemic colitis, or colitis of unknown origin.
* Fasting blood glucose > 6.9 mmol/l
* HbA1C > 6%
* Long QT, congenital or acquired
* Active pneumonitis
* Patients who require daily supplemental oxygen
* Inadequate renal function defined as creatinine clearance or radioisotope GFR < 60ml/min/1.73 m²
* Inadequate liver function defined as:
* Total bilirubin > 2.0 x ULN or conjugated bilirubin > 2.0 x ULN for age, and
* SGPT (ALT) or SGOT (AST) ≥ 1.5 x ULN for age, and
* Serum albumin < 30 g/L
* Inadequate fasting LDL cholesterol > 4.2 mmol/l
* Deprived of freedom by an administrative or court order, or benefiting from a system of legal protection (tutorship, curatorship or safeguard of justice).
* Not covered by health insurance

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2019-02-14 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Occurrence of dose limiting toxicities | less than 24 hours
  The dose limiting toxicity (DLT) is defined as a Grade 3 or more AE using the National Cancer Institute (NCI).
  If two out of up to six participants at the same dose level experience a DLT as defined above, subsequent cohorts will be dosed at a lower level as illustrated in the flow-chart below. At least six evaluable participants are required to establish the MTD (Maximum tolerated dose) at a specific dose level for both combinations.

CONTACTS AND LOCATIONS:
Locations (18):
- France (18):
  - CHU d'Angers, Angers
  - CHU de Bordeaux - GH Pellegrin, Bordeaux
  - Chu Dijon Bourgogne, Dijon
  - Hôpital Raymond Poincaré (AP-HP), Garches
  - Hôpital Jeanne de Flandre, Lille
  - HCL - Hôpital femme-mère-enfant, Lyon
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Hôpital Saint Eloi, Montpellier
  - CHU Hôtel Dieu, Nantes
  - CHU de Nice - Hôpital l'Archet 2, Nice
  - Hôpital Necker-Enfants malades, Paris
  - Hôpital Sud, Rennes
  - CHU La Réunion - Site GHSR, Saint-Pierre
  - CHU de Saint-Etienne Hôpital Nord, Saint-Priest-en-Jarez
  - Hôpital Larrey, Toulouse
  - Hôpital Trousseau, Tours
  - CHU de Nancy - Hôpital de Brabois, Vandœuvre-lès-Nancy
  - CHU de Nancy, Vandœuvre-lès-Nancy

REFERENCES:
- [Result] Luu M, Vabres P, Devilliers H, Loffroy R, Phan A, Martin L, Morice-Picard F, Petit F, Willems M, Bessis D, Jacquemont ML, Maruani A, Chiaverini C, Mirault T, Clayton-Smith J, Carpentier M, Fleck C, Maurer A, Yousfi M, Parker VER, Semple RK, Bardou M, Faivre L. Safety and efficacy of low-dose PI3K inhibitor taselisib in adult patients with CLOVES and Klippel-Trenaunay syndrome (KTS): the TOTEM trial, a phase 1/2 multicenter, open-label, single-arm study. Genet Med. 2021 Dec;23(12):2433-2442. doi: 10.1038/s41436-021-01290-y. Epub 2021 Aug 12. PMID 34385668